CLINICAL TRIAL: NCT06849115
Title: Effects of L-Carnitine in Amyotrophic Lateral Sclerosis Patients With CHCHD10 Mutations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ChaodongWang (Other)
Responsible Party: Sponsor-Investigator, ChaodongWang, Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALS-L-carnitine
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-02

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis; L-carnitine; CHCHD10; flail arm syndrome
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- L-carnitine group (Experimental)
  Interventions: Drug: L-Carnitine Injection，1000mg once daily

INTERVENTIONS:
Drug: L-Carnitine Injection，1000mg once daily — All patients were given L-carnitine therapy administered every 8 weeks, consisting of 1g L-carnitine diluted in 500 mL of 0.9% sodium chloride solution via intravenous infusion once daily. Each treatment cycle lasted 2 weeks, repeated at 8-week intervals for a total of 3 cycles, with L-carnitine 1g is administered orally once daily during the intervals between intravenous therapies.

SUMMARY:
The study was designed as a single-center, open-label, single-arm pilot study to estimate the safety and efficacy L-carnitine in ALS patients with CHCHD10 mutations.

DETAILED DESCRIPTION:
The study was designed as a single-center, open-label, single-arm pilot study and was performed at the ALS inpatient clinic of the Xuanwu Hospital in Beijing, China. ALS patients with CHCHD10 mutations were recruited to participate in the clinical trial. The patients were given L-carnitine therapy administered every 8 weeks, consisting of 1g L-carnitine diluted in 500 mL of 0.9% sodium chloride solution via intravenous infusion once daily. Each treatment cycle lasted 2 weeks, repeated at 8-week intervals for a total of 3 cycles, with L-carnitine 1g is administered orally once daily during the intervals between intravenous therapies. Primary end point was the changes of ALS-FRS-R scores, and secondary end points were the changes of plasm NfL level, FVC%, weight and ALSAQ-40 scores. Eligible patients were assessed at baseline and after 2, 10, 12, 20 and 30 weeks. At each visit, a detailed neurological examination, including assessment of general nerve function as well as quantitative and qualitative evaluation of the motor system, were performed for the patients. All adverse events (AEs) encountered and any serious events were to be recorded as true. Severity was graded according to the modified WHO criteria for toxicity (http://www.regsource. com/_Adverse_Event_Reporting/_adverse_event_ reporting.html) where applicable.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-80 years old
* ALS diagnosed as definite or probable as defined by the World Federation of Neurology revised El Escorial criteria
* Carrying pathogenic CHCHD10 mutations
* Capable of providing informed consent and following trial procedures
* Forced Vital Capacity (FVC) >40% of predicted value for gender, height, and age at the Screening Visit
* Subjects develop at less moderate degree of motor dysfunction, with ALS-FRS-R total scores less than 46
* Both male and female patients must agree to use adequate birth control for the whole duration of the study within 30 weeks
* Subjects are willing and expected to complete the 30-week follow up, including 3 times hospitalization.

Exclusion Criteria:

* Presence of tracheostomy
* History of known allergy to L-carnitine
* Abnormal liver function defined as AST and/or ALT > 3 times the upper limit of the normal
* Renal insufficiency as defined by eGFR < 60 mL/min/1.73m2
* Pregnant women or women currently breastfeeding
* Clinically significant unstable medical condition (other than ALS) that would pose a risk to the subject if they were to participate in the study
* Anything that, in the opinion of the Site Investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Changes of ALS-FRS-R scores | Eligible patients were assessed at baseline and after 2, 10, 12, 20 and 30 weeks.
  ALS-Functional Rating Scale-Revised (ALS-FRS-R) score ranges from 0 to 48, with higher scores indicating better motor function (0 = complete loss of motor function; 48 = intact/normal motor function)

SECONDARY OUTCOMES:
Changes of plasm NfL level | Eligible patients were assessed at baseline and after 10, 20 and 30 weeks.
Changes of FVC% | Eligible patients were assessed at baseline and after 10, 20 and 30 weeks.
  Predicted forced vital capacity (FVC)%
Changes of Weight | Eligible patients were assessed at baseline and after 2, 10, 12, 20 and 30 weeks.
Changes of ALSAQ-40 scores | Eligible patients were assessed at baseline and after 2, 10, 12, 20 and 30 weeks.
  The Amyotrophic Lateral Sclerosis Assessment Questionnaire-40 (ALSAQ-40) total scores range from 0 to 120. Higher scores indicate greater disease burden or poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China, China

IPD SHARING:
Plan to Share IPD: No